CLINICAL TRIAL: NCT03402841
Title: A Phase IIIb, Single-arm, Open-label Multicentre Study of Olaparib Maintenance Monotherapy in Platinum Sensitive Relapsed Non-Germline BRCA Mutated Ovarian Cancer Patients Who Are in Complete or Partial Response Following Platinum Based Chemotherapy
Brief Title: Multicentre Study of Olaparib Maintenance Monotherapy in Platinum Sensitive Relapsed Non gBRCAm Ovarian Cancer Patients
Acronym: OPINION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Myriad Genetics, Inc. (Industry); Covance (Industry); Theradex (Industry); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0816C00020; 2017-002767-17 (EudraCT Number)
Record Dates: First submitted 2018-01-03; First posted 2018-01-18 (Actual); Results first posted 2021-10-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Non-Germline BRCA Mutated Ovarian Cancer
Keywords: Ovarian cancer; non-gBRCA; Platinum; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: Single arm study
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Olaparib will be supplied as film-coated tablets containing 150 mg or 100 mg of olaparib.
  Patients will be administered olaparib orally twice daily (bid) at 300 mg.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — 300 mg twice daily - oral
  Other Names: Lynparza

SUMMARY:
The purpose of the study is to assess the efficacy and safety of single-agent olaparib as a maintenance treatment in patients with relapsed High Grade Serous Ovarian Cancer (including patients with primary peritoneal and/or fallopian tube cancer) or high grade endometrioid cancer who do not have known deleterious or suspected deleterious germline BRCA mutations (non-gBRCAm) and who had responded following platinum based chemotherapy

DETAILED DESCRIPTION:
Maintenance monotherapy with the potent polyadenosine 5'diphosphoribose [Poly (ADP-ribose)] polymerisation (PARP) inhibitor (PARPi) olaparib will significantly prolong progression-free survival (PFS) in platinum sensitive relapsed non-germline breast cancer susceptibility gene (BRCA) mutated ovarian cancer patients who are in complete or partial response following platinum based chemotherapy.

Olaparib is a potent PARPi (PARP-1, -2 and -3) that is being developed as an oral therapy, both as a monotherapy (including maintenance) and for combination with chemotherapy and other anticancer agents. PARP inhibition is a novel approach to targeting tumours with deficiencies in DNA repair mechanisms. PARP enzymes are essential for repairing DNA single strand breaks (SSBs). Inhibiting PARP enzymes leads to the persistence of SSBs, which are then converted to the more serious DNA double strand breaks (DSBs) during the process of DNA replication. During the process of cell division, DSBs can be efficiently repaired in normal cells by homologous recombination (HR) repair. Tumours with HR deficiencies (HRDs), such as ovarian cancers in patients with BRCA1/2 mutations, cannot accurately repair the DNA damage, which may become lethal to cells as it accumulates. In such tumour types, olaparib may offer a potentially efficacious and less toxic cancer treatment compared with currently available chemotherapy regimens.

While multiple randomized controlled trials (RCTs) have demonstrated that platinum sensitive BRCAm patients have profound response to maintenance treatment with PARP inhibitors, PARP inhibitors target cells with homologous recombination deficiency (HRD), of which BRCA mutation is only one type. Consistent with the mechanism of action of PARP inhibition, response has also been seen in multiple RCTs in patients who are platinum sensitive but whose tumours do not harbor BRCA mutations. Presumably these responders have defects in other components of HRR pathways, though currently available diagnostic technology is not adequate to reliably identify the full spectrum of HRR deficiencies. Instead, these data support the hypothesis that platinum sensitivity itself is a clinical selection factor for HRD.

ELIGIBILITY:
Key Inclusion Criteria:

* Female patients with histologically diagnosed relapsed HGSOC (including primary peritoneal and / or fallopian tube cancer) or high grade endometrioid ovarian cancer
* Documented gBRCA1/2 mutation status
* Patients must have completed at least 2 previous courses of platinum containing therapy
* Patients must have normal organ and bone marrow function measured within 28 days of starting study treatment
* ECOG performance status 0-1 (see Appendix E)
* Patients must have a life expectancy ≥16 weeks
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for repeated assessment OR No evidence of disease following a complete response to chemotherapy
* An appropriately prepared tumour sample from the cancer, of sufficient quantity and quality (as specified in the Central Laboratory Services Manual) must be available for future central testing of tumour genetic status

Exclusion Criteria:

* Patients receiving any systemic hormonal therapy, chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to start of study treatment
* Any previous treatment with PARP inhibitor, including olaparib
* Patients with a germline BRCA mutation that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental / lead to loss of function)
* Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
* Concomitant use of known strong CYP3A inhibitors and strong (or moderate CYP3A inducers
* Persistent toxicities (≥ Grade 2 Common Terminology Criteria for Adverse Event (CTCAE) adverse event) caused by previous cancer therapy, excluding alopecia
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML
* Patients with symptomatic uncontrolled brain metastases

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 279 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wilks, Study Director — AstraZeneca
Locations (82):
- Austria (4):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Vienna
  - Research Site, Wein
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Loverval
  - Research Site, Namur
  - Research Site, Wilrijk
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (6):
  - Research Site, Victoria, British Columbia
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Nový Jičín
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Denmark (2):
  - Research Site, Aalborg
  - Research Site, Aarhus
- Finland (3):
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Tampere
- Israel (6):
  - Research Site, Afula
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Ramat Gan
- Italy (6):
  - Research Site, Ancona
  - Research Site, Brescia
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Torino
- Netherlands (2):
  - Research Site, Breda
  - Research Site, Tilburg
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Poland (6):
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Portugal (2):
  - Research Site, Coimbra
  - Research Site, Lisbon
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Research Site, Ljubljana, Slovenia
- Spain (10):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Linköping
  - Research Site, Lund
- Switzerland (7):
  - Research Site, Basel
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Frauenfeld
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Zurich
- United Kingdom (9):
  - Research Site, Aberdeen
  - Research Site, Colchester
  - Research Site, Exeter
  - Research Site, Leeds
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Scarborough

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Background] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- [Background] Rottenberg S, Jaspers JE, Kersbergen A, van der Burg E, Nygren AO, Zander SA, Derksen PW, de Bruin M, Zevenhoven J, Lau A, Boulter R, Cranston A, O'Connor MJ, Martin NM, Borst P, Jonkers J. High sensitivity of BRCA1-deficient mammary tumors to the PARP inhibitor AZD2281 alone and in combination with platinum drugs. Proc Natl Acad Sci U S A. 2008 Nov 4;105(44):17079-84. doi: 10.1073/pnas.0806092105. Epub 2008 Oct 29. PMID 18971340
- [Background] Murai J, Huang SY, Das BB, Renaud A, Zhang Y, Doroshow JH, Ji J, Takeda S, Pommier Y. Trapping of PARP1 and PARP2 by Clinical PARP Inhibitors. Cancer Res. 2012 Nov 1;72(21):5588-99. doi: 10.1158/0008-5472.CAN-12-2753. PMID 23118055
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Helleday T. The underlying mechanism for the PARP and BRCA synthetic lethality: clearing up the misunderstandings. Mol Oncol. 2011 Aug;5(4):387-93. doi: 10.1016/j.molonc.2011.07.001. Epub 2011 Jul 22. PMID 21821475
- [Background] Hay T, Matthews JR, Pietzka L, Lau A, Cranston A, Nygren AO, Douglas-Jones A, Smith GC, Martin NM, O'Connor M, Clarke AR. Poly(ADP-ribose) polymerase-1 inhibitor treatment regresses autochthonous Brca2/p53-mutant mammary tumors in vivo and delays tumor relapse in combination with carboplatin. Cancer Res. 2009 May 1;69(9):3850-5. doi: 10.1158/0008-5472.CAN-08-2388. Epub 2009 Apr 21. PMID 19383921
- [Background] Ledermann J, Harter P, Gourley C, Friedlander M, Vergote I, Rustin G, Scott C, Meier W, Shapira-Frommer R, Safra T, Matei D, Macpherson E, Watkins C, Carmichael J, Matulonis U. Olaparib maintenance therapy in platinum-sensitive relapsed ovarian cancer. N Engl J Med. 2012 Apr 12;366(15):1382-92. doi: 10.1056/NEJMoa1105535. Epub 2012 Mar 27. PMID 22452356
- [Background] Pujade-Lauraine E, Ledermann JA, Selle F, Gebski V, Penson RT, Oza AM, Korach J, Huzarski T, Poveda A, Pignata S, Friedlander M, Colombo N, Harter P, Fujiwara K, Ray-Coquard I, Banerjee S, Liu J, Lowe ES, Bloomfield R, Pautier P; SOLO2/ENGOT-Ov21 investigators. Olaparib tablets as maintenance therapy in patients with platinum-sensitive, relapsed ovarian cancer and a BRCA1/2 mutation (SOLO2/ENGOT-Ov21): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1274-1284. doi: 10.1016/S1470-2045(17)30469-2. Epub 2017 Jul 25. PMID 28754483
- [Derived] Barnicle A, Ray-Coquard I, Rouleau E, Cadoo K, Simpkins F, Aghajanian C, Leary A, Poveda A, Lheureux S, Pujade-Lauraine E, You B, Ledermann J, Matulonis U, Gourley C, Timms KM, Lai Z, Hodgson DR, Elks CE, Dearden S, Egile C, Lao-Sirieix P, Harrington EA, Brown JS. Patterns of genomic instability in > 2000 patients with ovarian cancer across six clinical trials evaluating olaparib. Genome Med. 2024 Dec 18;16(1):145. doi: 10.1186/s13073-024-01413-5. PMID 39695768
- [Derived] Poveda A, Lheureux S, Colombo N, Cibula D, Lindemann K, Weberpals J, Bjurberg M, Oaknin A, Sikorska M, Gonzalez-Martin A, Madry R, Perez MJR, Ledermann J, Davidson R, Blakeley C, Bennett J, Barnicle A, Skof E. Olaparib maintenance monotherapy in platinum-sensitive relapsed ovarian cancer patients without a germline BRCA1/BRCA2 mutation: OPINION primary analysis. Gynecol Oncol. 2022 Mar;164(3):498-504. doi: 10.1016/j.ygyno.2021.12.025. Epub 2022 Jan 19. PMID 35063276
- [Derived] Poveda AM, Davidson R, Blakeley C, Milner A. Olaparib maintenance monotherapy in platinum-sensitive, relapsed ovarian cancer without germline BRCA mutations: OPINION Phase IIIb study design. Future Oncol. 2019 Nov;15(32):3651-3663. doi: 10.2217/fon-2019-0343. Epub 2019 Sep 25. PMID 31553234
- See also: D0816C00020 CSP-v-3_Final Draft_13Sep21_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00020&attachmentIdentifier=486daa20-bd4a-47b0-bc50-4a91568f722f&fileName=d0816c00020-csp-v-3_Final_Draft_13Sep21_Redacted.pdf&versionIdentifier=
- See also: D0816C00020-sap-v-2_Final_Draft_13Sep21_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00020&attachmentIdentifier=481a4401-0306-4d17-a5fc-edfdd6258606&fileName=d0816c00020-sap-v-2_Final_Draft_13Sep21_Redacted.pdf&versionIdentifier=
- See also: D0816C00020-study-synopsis-pa_Final draft_13Sep21_Redacted.pdf — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00020&attachmentIdentifier=9826555e-52bc-47f7-9750-58a3f471bb4a&fileName=d0816c00020-study-synopsis-pa_Final_Draft_13Sep21_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D0816C00020&attachmentIdentifier=597429d8-3f37-49d5-bd20-89cdcf0edd1d&fileName=D0816C00020_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIIb, single-arm, open-label multicentre study to assess the efficacy and safety of single-agent olaparib as a maintenance treatment in eligible patients. A total of 279 patients from 17 countries were enrolled in this study.
Pre-assignment Details: Olaparib was administered to all patients at a starting dose of 300 milligrams (mg) twice daily. Dose reductions were required in patients experiencing toxicities or due to concomitant medication (CM).
Groups:
- Olaparib: Olaparib was administered to all patients at a starting dose of 300 mg twice daily. Dose reductions were required in patients experiencing toxicities or due to CM.
  Patients continued with olaparib until documented disease progression as assessed by the Investigator or unacceptable toxicity or for as long as they did not meet any other discontinuation criteria.
Period: Overall Study
Arm/Group | Olaparib
Started | 279
Completed | 128
Not Completed | 151
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Death | 146

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all enrolled patients assigned to olaparib.
Arm/Group | Olaparib
Number analyzed (Participants) | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.19)
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 22
  >=50 - <65 years | 110
  >=65 - <75 years | 113
  >=75 years | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 273
  Black or African American | 1
  Asian | 2
  Unspecified | 2
  Missing | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 271
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of first dose until the date of objective radiological disease progression. Assessed according to modified Response Evaluation Criteria In Solid Tumours Version 1.1 (RECIST 1.1) or death (by any cause in the absence of progression). Progression was determined by investigator assessment, RECIST 1.1. Calculated using the Kaplan-Meier technique. Confidence intervals (CI) for median PFS was derived based on Brookmeyer-Crowley method.
Time Frame: Up to maximum of 32 months
Population: The FAS included all enrolled patients assigned to olaparib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 279
months | 9.2 [7.6 to 10.9]

2. Secondary Outcome: Time to First Subsequent Therapy or Death (TFST)
Description: TFST is defined as the time from date of first dose to date of first subsequent treatment commencement or death due to any cause if this occurs before commencement of first subsequent treatment. Calculated using the Kaplan-Meier technique. CI for median TFST was derived based on Brookmeyer-Crowley method.
Time Frame: Up to a maximum of 43 months
Population: The FAS included all enrolled patients assigned to olaparib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 279
months | 13.9 [11.5 to 16.6]

3. Secondary Outcome: Time to Treatment Discontinuation or Death (TDT)
Description: TDT is defined as the time from date of first dose to date of study drug discontinuation or death due to any cause if this occurs before study drug discontinuation. Calculated using the Kaplan-Meier technique. CI for median TDT was derived based on Brookmeyer-Crowley method.
Time Frame: Up to a maximum of 43 months
Population: The FAS included all enrolled patients assigned to olaparib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 279
months | 9.6 [7.8 to 11.1]

4. Secondary Outcome: PFS by Homologous Recombination Deficiency (HRD)/ Breast Cancer Susceptibility Gene Mutation (Mutated) (BRCAm) Status
Description: HRD/BRCAm status was based on the central blood and tumour assessments. Assessed according to modified RECIST 1.1 or death (by any cause in the absence of progression). Progression was determined by investigator assessment, RECIST 1.1. Calculated using the Kaplan-Meier technique. CI for median PFS was derived based on Brookmeyer-Crowley method.
Time Frame: Up to maximum of 32 months
Population: The FAS included all enrolled patients assigned to Olaparib. Only FAS patients with available central assessment are reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 242
months
  HRD status positive and/or sBRCAm subgroup: number analyzed (Participants) | 121
  HRD status positive and/or sBRCAm subgroup | 11.1 [9.2 to 14.6]
  HRD status positive, non-BRCAm subgroup: number analyzed (Participants) | 94
  HRD status positive, non-BRCAm subgroup | 9.7 [8.1 to 13.6]
  HRD status negative subgroup: number analyzed (Participants) | 115
  HRD status negative subgroup | 7.3 [5.5 to 9.0]
  sBRCAm subgroup: number analyzed (Participants) | 27
  sBRCAm subgroup | 16.4 [12.8 to NA] — The upper CI was not calculable due to insufficient progression events.
  gBRCAm subgroup: number analyzed (Participants) | 6
  gBRCAm subgroup | 12.1 [3.7 to NA] — The upper CI was not calculable due to insufficient progression events.

5. Secondary Outcome: Chemotherapy-free Interval (CT-FI)
Description: CT-FI is defined as the time from the date of the last dose of platinum chemotherapy prior to olaparib maintenance therapy until the date of initiation of the next anticancer therapy. Calculated using the Kaplan-Meier technique. CI for median CT-FI was derived based on Brookmeyer-Crowley method.
Time Frame: Up to a maximum of 43 months
Population: The FAS included all enrolled patients assigned to olaparib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 279
months | 17.9 [13.8 to 23.3]

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of olaparib to the date of death from any cause. Calculated using the Kaplan-Meier technique. CI for median OS was derived based on Brookmeyer-Crowley method.
Time Frame: Up to a maximum of 43 months
Population: The FAS included all enrolled patients assigned to olaparib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Olaparib
Number analyzed (Participants) | 279
months | 32.7 [29.5 to 35.3]

7. Secondary Outcome: Percentage of Patients With Any Improvement From Baseline in Trial Outcome Index (TOI) Score at Any Point During the Treatment Period
Description: Improvement was defined as a functional assessment of cancer therapy - ovarian (FACT-O) TOI response of "any improvement" at any time point over the course of treatment. The TOI is an established single targeted index composed of the following scales of the FACT-O: physical and functional well-being and additional concerns. The range of possible scores for the FACT-O TOI is 0-100, with a higher score indicating better health related quality of life (HRQoL). An increase in score from baseline indicates an improvement in HRQoL.
Time Frame: Baseline up to a maximum of 32 months
Population: The FACT-O set consisted of all FAS patients with at least a baseline and a post-baseline assessment (excluding the end of treatment and 30-day follow up assessments).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Olaparib
Number analyzed (Participants) | 249
percentage of patients | 64.3 [58.0 to 70.2]

8. Secondary Outcome: Percentage of Patients With a 10-Point Deterioration From Baseline in TOI Score at Any Point During the Treatment Period
Description: 10-point deterioration was defined as a FACT-O TOI response of "10-point deterioration" at any time point over the course of treatment. The TOI is an established single targeted index composed of the following scales of the FACT-O: physical and functional well-being and additional concerns. The range of possible scores for the FACT-O TOI is 0-100, with a higher score indicating better HRQoL. A decrease in score of at least 10 points from baseline was defined as a clinically meaningful deterioration.
Time Frame: Baseline up to a maximum of 32 months
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Olaparib
Number analyzed (Participants) | 249
percentage of patients | 42.6 [36.3 to 49.0]

ADVERSE EVENTS:
Time Frame: Includes adverse events with an onset date on or after the date of first dose and up to and including 30 days following the date of last dose of olaparib, up to a maximum of 43 months
Description: Safety Analysis set consisted of all patients in the FAS who received at least 1 dose of olaparib.
Groups:
- Olaparib 300mg BID: Olaparib was administered to all patients at a starting dose of 300 mg twice daily. Dose reductions were required in patients experiencing toxicities or due to CM.
  Patients continued with olaparib until documented disease progression as assessed by the Investigator or unacceptable toxicity or for as long as they did not meet any other discontinuation criteria.
Arm/Group | Olaparib 300mg BID
All-Cause Mortality (participants affected / at risk) | 146/279
Serious Adverse Events (participants affected / at risk) | 58/279
Other Adverse Events (participants affected / at risk) | 268/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg BID (N=279)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Biliary dyskinesia (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 22 (31)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic embolus (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300mg BID (N=279)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (31)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 16 (23)
Swelling (General disorders) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Atypical mycobacterial lower respiratory tract infection (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4)
Covid-19 (Infections and infestations) | 2 (2)
Candida infection (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 3 (3)
Arrhythmia (Cardiac disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Conjunctivitis viral (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 10 (15)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 2 (2)
Enteritis infectious (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 6 (7)
Laryngitis (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Nail infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 15 (17)
Oral candidiasis (Infections and infestations) | 3 (3)
Oral herpes (Infections and infestations) | 1 (3)
Otitis media (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Tachycardia (Cardiac disorders) | 2 (2)
Pneumonia viral (Infections and infestations) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2)
Salmonellosis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 12 (12)
Urethritis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 27 (36)
Viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Hand fracture (Injury, poisoning and procedural complications) | 2 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (8)
Amylase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (9)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (6)
Blood creatine increased (Investigations) | 3 (4)
Blood creatinine increased (Investigations) | 29 (46)
Blood potassium decreased (Investigations) | 1 (2)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 4 (4)
Creatinine renal clearance decreased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 102 (197)
Vertigo (Ear and labyrinth disorders) | 4 (5)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (6)
Mean cell volume increased (Investigations) | 2 (2)
Monocyte count increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 14 (32)
Occult blood (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 16 (33)
Sars-cov-2 test positive (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2)
Troponin i increased (Investigations) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1)
Vitamin b12 decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 6 (6)
Weight increased (Investigations) | 3 (3)
White blood cell count decreased (Investigations) | 13 (29)
Decreased appetite (Metabolism and nutrition disorders) | 32 (34)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Amaurosis fugax (Eye disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 13 (20)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (6)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (30)
Cataract (Eye disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (30)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (8)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (16)
Dry eye (Eye disorders) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (11)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Eye disorder (Eye disorders) | 1 (1)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vision blurred (Eye disorders) | 2 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1)
Amnesia (Nervous system disorders) | 1 (2)
Balance disorder (Nervous system disorders) | 1 (3)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 17 (22)
Dysgeusia (Nervous system disorders) | 40 (44)
Dyskinesia (Nervous system disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 24 (27)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Neurotoxicity (Nervous system disorders) | 4 (4)
Paraesthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Polyneuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 3 (4)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Trigeminal nerve disorder (Nervous system disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 13 (13)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (6)
Bradyphrenia (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 7 (7)
Genito-pelvic pain/penetration disorder (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 14 (14)
Irritability (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1)
Tension (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 9 (10)
Haematuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 3 (3)
Polyuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 3 (4)
Urinary tract disorder (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 43 (52)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 5 (5)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (36)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 6 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 16 (18)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (16)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1)
Aerophagia (Gastrointestinal disorders) | 2 (3)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 10 (13)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Angular cheilitis (Gastrointestinal disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Embolism (Vascular disorders) | 2 (2)
Flushing (Vascular disorders) | 4 (5)
Haematoma (Vascular disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Hot flush (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 7 (7)
Hypotension (Vascular disorders) | 2 (4)
Lymphoedema (Vascular disorders) | 2 (2)
Peripheral coldness (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Erythropenia (Blood and lymphatic system disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 23 (28)
Defaecation urgency (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 40 (55)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 16 (18)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 15 (25)
Eructation (Gastrointestinal disorders) | 1 (1)
Faecal vomiting (Gastrointestinal disorders) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 8 (8)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 136 (187)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 6 (9)
Oral mucosal exfoliation (Gastrointestinal disorders) | 1 (1)
Palatal disorder (Gastrointestinal disorders) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 13 (13)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 45 (68)
Adhesion (General disorders) | 1 (1)
Asthenia (General disorders) | 46 (57)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 4 (4)
Chills (General disorders) | 2 (2)
Early satiety (General disorders) | 2 (2)
Face oedema (General disorders) | 2 (2)
Fatigue (General disorders) | 82 (103)
Neutropenia (Blood and lymphatic system disorders) | 31 (62)
Inflammation (General disorders) | 1 (1)
Influenza like illness (General disorders) | 5 (5)
Infusion site extravasation (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Mass (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 9 (10)
Non-cardiac chest pain (General disorders) | 5 (5)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 13 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT03402841/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03402841/SAP_003.pdf